CLINICAL TRIAL: NCT02292498
Title: Thermal Imaging to Diagnose and Monitor Suspected Bacterial Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Patricia L. Hibberd, Chief, Division of Pediatric Global Health, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2014P001327
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Infections, Bacterial; Pneumonia, Bacterial
Keywords: imaging, diagnostic; feasibility
MeSH Terms: conditions — Bacterial Infections; Pneumonia, Bacterial; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FLIR ONE thermal camera (Experimental): Thermal camera (FLIR ONE)
  Interventions: Device: FLIR ONE

INTERVENTIONS:
Device: FLIR ONE

SUMMARY:
The purpose of this study is to test the feasibility of using thermal images to diagnose bacterial pneumonia instead of a chest x-ray in the future. More specifically, the objectives of this study are: 1) to determine if thermal imaging, using a commercial thermal camera can detect areas of heat emitted from the chest in similar locations to where a chest X-ray shows focal consolidation consistent with bacterial pneumonia; 2) to evaluate whether changes in heat emitted from the chest changes over time if it is possible to obtain serial images of the chest.

ELIGIBILITY:
Inclusion Criteria:

* Subject sent for a clinical chest X-ray (not research) to rule out pneumonia
* Thermal images obtained using FLIR ONE within 4 hours of the chest x-ray
* Signed informed consent obtained
* Subject is a patient at a participating clinic at Massachusetts General Hospital

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
feasibility of diagnosis of bacterial pneumonia | 4 hours
  Thermal imaging will be compared to the chest x-ray taken within 4 hours to see if bacterial pneumonia is present

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L Hibberd, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No